CLINICAL TRIAL: NCT05089552
Title: Psychiatric Assessment and Quality of Life of Family Caregivers of Addicts
Brief Title: Quality of Life of Caregivers of Addicts
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Saleh Sharkawy, principal investigator, Assiut University
Other Study IDs: qolfc
Record Dates: First submitted 2021-10-10; First posted 2021-10-22 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Addiction
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 1-WHOQOL-BREF(WHO-Quality of life-BREFF) Arabic version Scale — WHOQOL-BREF(WHO-Quality of life-BREFF) Arabic version Scale The WHOQOL-BREF is composed of 26 self-administered items. Using a 5-point Likert response scale ranging from 1 (very dissatisfied/very poor) to 5 (very satisfied/very good), family caregivers were asked to rank each item accordingly. Caregivers were asked to respond to the items indicating their assessment of QOL during the preceding 2 weeks, Ohaeri and Awadalla developed and tested the Arabic version of the WHOQOL-BREF among an Arab population in Kuwait. The translated Arabic WHOQOL-BREF has considerable reliability and validity indices . As reported in the Kuwaiti study, a satisfactory (≥0.7) Cronbach's alpha was reported for the full questionnaire and the domains
Other: SCL-90-R(Symptoms Checklist-90-Revised) Arabic version scale — developed by Derogatis et al. and El-Behairy. established the validity and reliability of the Arabic version.SCL-90-R is a 90-item self-report symptom inventory, and reflect the psychologic symptom pattern of psychiatric and medical patients. Each item of the "90" is rated on a five-point scale of distress (0-4), ranging from "not at all" to "extremely".Under usual circumstances, SCL-90-R requires between 12 and 15 minutes to be completed.SCL-90-R is a measure of the current psychologic symptom status. It is not a measure of personality, except indirectly, in that certain personality disorders may manifest a characteristic profile on the primary symptom dimensions.
Other: addiction severity index — a semi-structured interview that takes approximately 45 minute. developed to evaluate treatment outcome in substance abusers. The instrument focuses on seven areas that are typically affected in the lives of substance abusers: medical status, employment, drug use, alcohol use, legal status, family/social status, and psychiatric status. Information regarding frequency, duration, and severity of problems in these seven areas is collected for both lifetime and recent (past 30 days) history. The ASI provides two types of scores: severity and subjective ratings of the client's need for treatment, and composite scores of problem severity during the prior 30 days. Specific alcohol-related questions include total lifetime years of use, money spent on alcohol, and number of days that alcohol problems are experienced.

SUMMARY:
American Society of Addiction Medicine defined Addiction as a treatable, chronic medical disease involving complex interactions among brain circuits, genetics, the environment, and an individual's life experiences. People with addiction use substances or engage in behaviors that become compulsive and often continue despite harmful consequences.

Addiction is considered as a "family disease." Addiction affects the individual as well as those around them in terms of occupational and social dysfunction, physical and emotional distress, and financial burden which has a serious impact on the lives of the significant others.

DETAILED DESCRIPTION:
Addiction is a multifaceted problem- it negatively alters the quality of life of not only addicts but also the family members who live with them. Caregiving to an individual suffering from addiction is physically, mentally, socially and emotionally challenging. These caregivers are most burdened as the assistance they provide is multidimensional.

The Quality of Life Group of the World Health Organization (WHO) Division of Mental Health has defined QOL as "an individual's perception of their position in life in the context of the culture and value system in which they live and in relation to their goals, expectations, standards, and concerns " .

Family members are not all equally affected and they suffer in different degrees based on their closeness to the addict and distance from the addict's behavior. Most of the time, a member of the family assumes the role of caregiver, and he or she is most burdened from this process.

The Family Caregiver Alliance (2014) defines family (or informal) caregivers as "any relative, partner, friend, or neighbor who has a significant personal relationship with, and provides a broad range of assistance for, an older person or an adult with a chronic or disabling condition" .

Researchers have described addiction as one of the significant causes of family destruction and disturbed relationship.Family relationships are at risk owing to addiction and associated hazards. Researches addressing the health issues of families have reported numerous mental health problems among children and spouses of addicts. A study has depicted children of addict fathers experiencing depression, anxiety and hypomania. Children of addicts also suffered from different internalised and externalised problem in men.

However, published studies on family caregivers of addicts are limited. This study aimed to evaluate QOL and psychiatric symptoms in family caregivers of addicts.

ELIGIBILITY:
Inclusion Criteria:

* As defined by The Family Caregiver Alliance (2014) "any relative, partner, friend, or neighbor who has a significant personal relationship with, and provides a broad range of assistance for, an older person or an adult with a chronic or disabling condition" .
* aged ≥18 years old.
* being a family caregiver for more than three months (considered the minimum time for the caregivers to be able to feel the effects of care).
* living or residing near the drug-dependent.

Exclusion Criteria:

* who stopped living in the city
* the presence of previous psychiatric illness and caregiver who was also addicts. • Refuse to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Family caregivers of addicts who come to an addiction clinic and unit of neuropsychiatry hospital of assiut university hospital
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
quality of life evaluation | 2 weeks
  evaluation of quality of life by WHO-QOL-BREFF scale
psychiatric symptoms | 12-15 minutes
  evaluation of psychiatric symptoms by Symptom Checklist-90-Revised (SCL-90-R)

CONTACTS AND LOCATIONS:
Overall Officials: Saleh Ahmed Mahmoud, Resident, Principal Investigator — Assiut University; ALaa EL-DIN Mohamed darweesh, MD, Study Chair — Assiut University; Mohamed Fawzy Mohamed, AP, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vaishnavi R, Karthik MS, Balakrishnan R, Sathianathan R. Caregiver Burden in Alcohol Dependence Syndrome. J Addict. 2017;2017:8934712. doi: 10.1155/2017/8934712. Epub 2017 May 21. PMID 28607798
- [Background] The World Health Organization Quality of Life assessment (WHOQOL): position paper from the World Health Organization. Soc Sci Med. 1995 Nov;41(10):1403-9. doi: 10.1016/0277-9536(95)00112-k. PMID 8560308
- [Background] Settley C. The physical and psychological wellbeing of caregivers of individuals suffering from substance addiction. Arch Psychiatr Nurs. 2020 Jun;34(3):107-109. doi: 10.1016/j.apnu.2020.03.007. Epub 2020 Mar 12. PMID 32513458
- [Background] Rafiq M, Sadiq R. Caregiver Stress, Perceived Stigma and Mental Health in Female Family Members of Drug Addicts: Correlational Study. J Pak Med Assoc. 2019 Sep;69(9):1300-1303. PMID 31511715